CLINICAL TRIAL: NCT05756595
Title: A Preliminary Clinical Study of Freshly Manufactured 35kDa Hyaluronan Fragment in the Treatment of Herpes Zoster Pain and Shoulder, Neck, Back and Temporal Pain
Brief Title: A Clinical Study of Freshly Manufactured 35kDa Hyaluronan Fragment in the Treatment of Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dove Medical Press Ltd (Network)
Collaborators: The Affiliated Hospital of Qingdao University (Other); Nakhia Impex LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: hui19590204
Record Dates: First submitted 2023-02-09; First posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-02

CONDITIONS: Shoulder Pain; Neck Pain; Back Pain; Temporal Pain; Herpes Zoster Pain
Keywords: hyaluronidase; Hyaluronan; 35kDa Hyaluronan fragment; pain caused by herpes zoster; pain caused by shoulder neck back and temporal
MeSH Terms: conditions — Shoulder Pain; Neck Pain; Back Pain

STUDY DESIGN:
Intervention Model Description: A self-controlled an open label clinical study(An investigator-initiated off-label use clinical study)
Masking Description: A self-controlled an open label clinical study(An investigator-initiated off-label use clinical study)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 35kDa hyaluronan fragment HA35 injection (Experimental): 100 mg Hyaluronan is locally injected at the pain point or where the nerve trunk is innervated by the pain point.
  Interventions: Drug: HA35(L20200708MP07707, Ministry of Health, Mongolia) was freshly manufactured by mixing hyaluronidase PH20 injectable solution (H31022111) and high-molecular-weight HA injectable solution (H20174089)

INTERVENTIONS:
Drug: HA35(L20200708MP07707, Ministry of Health, Mongolia) was freshly manufactured by mixing hyaluronidase PH20 injectable solution (H31022111) and high-molecular-weight HA injectable solution (H20174089) — This group will inject once a week. Evaluation of pain score after 30 seconds and 3 hours.
  Other Names: HA35

SUMMARY:
Local used high molecular weight Hyaluronan (HA) with high viscosity has a variety of receptors in the human body, including CD44, LYVE-1, RHAMM, HARE, Siglec-9, TLR2, CEMIP and TMEM2. Intra-articular local injection of HA has a certain degree of analgesic effect. Local injection of HA into the nerve trunk directed by ultrasound was used for the treatment of neuropathic pain. It was reported that the analgesic effect of HA is regulated by TRPV1 ion channels. This study hypothesizes that hyaluronidase cleaves HA to generate low molecular weight HA fragments HA35 with good tissue permeability, which may bind to a variety of HA receptors on the cell surface within the tissues and produce a broad-spectrum analgesic effect. In this study, 35kDa Hyaluronan fragment HA35 was prepared by mixing hyaluronidase PH20 injection and high molecular weight Hyaluronan (HA) injection at room temperature for 20 minutes. In this study, hyaluronidase injection and Hyaluronan injection were off-label used to conduct an investigator-initiated study (IIT or IIS) for the treatment of herpes zoster and shoulder, neck, back and temporal pain.

DETAILED DESCRIPTION:
Bioactive Hyaluronan fragment HA35 of 35kDa was isolated from human colostrum. Literature studies have shown that female breast hyaluronidase and male testicular sperm acrosomal hyaluronidase PH20 come from the same gene. The investigators, recombinant human hyaluronidase PH20 and neutral hyaluronidase (PH20 or SPAM1) of bovine testicular sperm acrosome were used to cleave macromolecular Hyaluronan. Regardless of the cutting time, the Hyaluronan fragment HA35 with an average molecular weight 35kDa was produced(Registration number L20200708MP07707, Ministry of Health, Mongolia). Hyaluronidase injection is often used to improve the penetration and absorption of other injectable drugs. Hyaluronidase injection is also used to degrade excessive use of cosmetic injection or improper use of cross-linked macromolecular Hyaluronan fillers, which is an off-label drug use of hyaluronidase（https://www.realself.com/news/ hyaluronidase-dissolve-fillers）. In this study, Hyaluronan fragment HA35 of 35kDa was prepared by mixing hyaluronidase injection extracted from bovine testis (hyaluronidase for injection, H31022111) and Hyaluronan injection (sodium hyaluronate injection, H20174089) at room temperature for 20 minutes. Its analgesic effect on herpes zoster, shoulder, neck, back, and temporal pain was studied.

In this study, off-label drug use of hyaluronidase injection and Hyaluronan injection （https://www.realself.com/news/ hyaluronidase-dissolve-fillers）were used in the clinical study of shoulder, neck, back and temporal pain and herpes zoster pain, namely investigator initiated trails. In this clinical trial, 26 patients with shoulder, neck, back and temporal pain were studied in the Department of pain diagnosis and treatment of the affiliated Hospital of Qingdao University. Ten patients with herpes zoster were treated in the pain Department of the affiliated Hospital of Qingdao University. According to the ratio of 100mg high molecular Hyaluronan / 2000 unit hyaluronidase, the high molecular Hyaluronan injection (sodium hyaluronate injection, H20174089) and the hyaluronidase injection extracted from bovine testis (hyaluronidase for injection) were mixed at room temperature for 20 minutes. Each time according to the amount of high molecular Hyaluronan containing 100 mg Hyaluronan and hyaluronidase mixture, pain point area and pain point area of the nerve trunk innervation of the local multi-point injection. Then, pain scale was used to evaluate and record the pain relief of patients before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Shoulder, neck, back and temporal pain. The course of the disease ranged from 0 to 8 months.
* Herpes zoster pain. The course of 0-2 months.

Exclusion Criteria:

* Individuals with severe spinal pathology (including fractures, inflammatory diseases and tumors)

Ages: 39 Years to 63 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2023-02-08 (Actual)

PRIMARY OUTCOMES:
Pain scores of all shoulder, neck, back, temporal and herpes zoster pain | 3 hours
  The pain scale is a tool that doctors use to help assess patients' pain. Each patient rated their pain on a scale of 0 to 10. 0 means "no pain" and 10 means "the most painful". Statistical t-test was used to calculate and evaluate the pain intensity, which was expressed as mean ±standard deviation.

CONTACTS AND LOCATIONS:
Locations (1):
- Qingdao University Affiliated Hospital, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: published precinical study and international granted patent
Access Criteria: Anti-Inflammatory Effects of the 35kDa Hyaluronic Acid Fragment (B-HA/HA35); APPLICATION OF LOW-MOLECULAR-WEIGHT HYALURONIC ACID(LMW-HA) FRAGMENTS(INJECTION) WO/2017/186088 US20200254005 EP3479830 AU2017255833 CA3049286
URL: http://www.dovepress.com/articles.php?article_id=80993；https://patentscope.wipo.int/search/en/detail.jsf?docId=CA249072967&_cid=P22-LDWT33-38680-1

REFERENCES:
- [Result] Jia X, Shi M, Wang Q, Hui J, Shofaro JH, Erkhembayar R, Hui M, Gao C, Gantumur MA. Anti-Inflammatory Effects of the 35kDa Hyaluronic Acid Fragment (B-HA/HA35). J Inflamm Res. 2023 Jan 13;16:209-224. doi: 10.2147/JIR.S393495. eCollection 2023. PMID 36686276
- [Result] APPLICATION OF LOW-MOLECULAR-WEIGHT HYALURONIC ACID(LMW-HA) FRAGMENTS(INJECTION) WO/2017/186088 US20200254005 EP3479830 AU2017255833 CA3049286
- See also: Related Info — http://patentscope.wipo.int/search/en/detail.jsf?docId=CA249072967&_cid=P22-LDWT33-38680-1